CLINICAL TRIAL: NCT02708875
Title: Microvascular Insulin Resistance and Mixed Meal Challenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menzies Institute for Medical Research (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Michelle Keske, Senior Research Fellow, Menzies Institute for Medical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: H14086
Record Dates: First submitted 2016-02-17; First posted 2016-03-15 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Insulin Resistance
Keywords: Microvascular; Insulin resistance; Mixed Meal; Glucose tolerance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mixed Meal Challenge (Experimental): Participants will consume a liquid mixed meal (~300 calories - fat, carbohydrate, and protein) for monitoring changes in glucose metabolism, plasma insulin and microvascular responses in skeletal muscle over 2 hours.
  Interventions: Other: Mixed Meal Challenge
- Glucose Challenge (Active Comparator): Participants will consume a glucose challenge (50g glucose) for monitoring changes in glucose metabolism, plasma insulin and microvascular responses in skeletal muscle over 2 hours.
  Interventions: Other: Glucose Challenge

INTERVENTIONS:
Other: Mixed Meal Challenge — Liquid mixed meal (300 calories - fat, carbohydrate, and protein).
  Arms: Mixed Meal Challenge
Other: Glucose Challenge — Glucose drink (50g glucose)
  Arms: Glucose Challenge

SUMMARY:
Insulin resistance (or pre-diabetes) is diagnosed using the oral glucose tolerance test. However, high blood glucose levels during this test may adversely impact on microvascular function. Investigators will determine whether a liquid mixed meal challenge (from carbohydrate, protein and fat) is a more appropriate test for assessing microvascular-derived insulin resistance.

DETAILED DESCRIPTION:
After consuming a meal, 80% of glucose is disposed in skeletal muscle. Our research group has demonstrated that microvascular blood flow in skeletal muscle plays an integral role in this process. Physiological doses of insulin stimulate microvascular blood flow, and that this increase is associated with enhanced glucose uptake by muscle. This microvascular action of insulin is lost during insulin resistance and type 2 diabetes.

The oral glucose tolerance test (GTT) is the gold standard for assessing insulin resistance and pre-diabetes and is used world-wide. However high blood glucose levels following a glucose load may adversely impact on microvascular function. The aim of this project is to determine whether a mixed meal challenge (liquid drink consisting of carbohydrate, fat and protein) is a better test for assessing microvascular-derived insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years.
* Normal to overweight (BMI 19-35 kg/m2).
* Normotensive (Seated brachial blood pressure <160/100 mmHg).
* Considered healthy (HbA1c <6.5 %) or have clinically diagnosed type 2 diabetes.
* Either have a parent with T2D, or no family history of type 2 diabetes for two generations.
* Have given signed informed consent to participate in the study

Exclusion Criteria:

* Age <18 yrs or >70 yrs
* Morbidly obese with a BMI ≥36 kg/m2
* History of myocardial infarction or stroke
* History of malignancy within past 5 years (except for non-melanoma skin cancers)
* Current smoker
* History of severe liver disease
* History of drug or alcohol abuse
* Elective major surgery during the course of the study
* Pregnancy/lactation
* Participation or intention to participate in another clinical research study during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in muscle microvascular blood flow | 1 hr
  Microvascular responses will be measured by contrast enhanced ultrasound before and 1hr after each challenge.

SECONDARY OUTCOMES:
Changes in blood glucose levels | 2 hr
  Blood glucose levels will be measured at 0, 15, 30, 60, 90 and 120 min following each challenge.
Changes in plasma insulin levels | 2hr
  Plasma insulin levels will be measured at 0, 15, 30, 60, 90 and 120 min following each challenge.
Changes in the respiratory exchange ratio (RER) | 1 hr
  Changes in RER will be measured by metabolic cart during each challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Keske, PhD, Principal Investigator — Menzies Institute for Medical Research
Locations (2):
- Australia (2):
  - Menzies Institute for Medical Research, Hobart, Tasmania
  - Deakin University, Burwood, Victoria

IPD SHARING:
Plan to Share IPD: No